CLINICAL TRIAL: NCT05324215
Title: Effects of Transversalis Fascia Plane Block and Rectus Sheath Block on Opioid Consumption in Renal Transplantation Donors
Brief Title: Transversalis Fascia Plane Block and Rectus Sheath Block in Renal Transplantation Donors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Koc University Hospital (Other)
Responsible Party: Principal Investigator, Özlem Özkalaycı, Principal Investigator, Koc University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Koc University Hospital
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversalis Fascia Plane Block and Rectus Sheath Block Group (Active Comparator): Transversalis Fascia Plane Block and Rectus Sheath Block will be administered to this group.
  Interventions: Procedure: Transversalis fascia plane block and rectus sheath block; Device: Intravenous fentanyl patient control device
- Control Group (Sham Comparator): No regional anesthesia technique will be applied to the control group.
  Interventions: Device: Intravenous fentanyl patient control device

INTERVENTIONS:
Procedure: Transversalis fascia plane block and rectus sheath block — Transversalis fascia plane block and rectus sheath block will be administered after the surgery.
  Arms: Transversalis Fascia Plane Block and Rectus Sheath Block Group
Device: Intravenous fentanyl patient control device — 24-hour fentanyl consumption will be recorded.

SUMMARY:
Transversalis fascia plane block (TFPB) is a relatively new, easy-to-apply and safe regional anesthesia technique used to provide postoperative analgesia in various surgeries. It has been shown that TFPB and rectus sheath block (RSB) administration reduces opioid consumption and related side effects in patients undergoing surgery with general anesthesia. To our knowledge, there is no study examining TFPB in donor nephrectomy.

The investigators aimed to prospectively examine the effect of TFPB and RSB on opioid consumption in postoperative period on donors who will undergo laparoscopic nephrectomy in renal transplantation surgery.

ELIGIBILITY:
Inclusion Criteria:

* Donor patients scheduled for elective nephrectomy in renal transplantation surgery
* American Society of Anesthesiologists (ASA) I-II
* Patients who are aged between 18-75

Exclusion Criteria:

* Skin infection at the block area
* Coagulation disorder and using anticoagulant drugs
* End-stage organ and system failure
* Severe pulmonary and/or cardiovascular problems
* Substance addiction or known psychiatric or mental problems
* Chronic painkiller usage

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-02-17 (Estimated); Study Completion 2023-02-17 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption retrieved from patient records | up to 24 hours
  the amount of fentanyl required by the patient and given by the device will be recorded for the first 24 hours.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) | up to 24 hours
  Pain of patients will be evaluated and recorded according to NRS. A NRS requires the patient to rate their pain on a defined scale between 0 and10 (0 is no pain and 10 is the worst pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Koç University Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No